CLINICAL TRIAL: NCT04332289
Title: Deciphering the Enigma of Postprandial Hyperinsulinaemic Hypoglycaemia After Bariatric Surgery, Part 1 A: Assessing Insulin Turnover Using an In-vivo Deuterated Water Experiment. A Proof-of-concept Study.
Brief Title: Assessing Insulin Turnover Using an In-vivo Deuterated Water Experiment.
Acronym: DEEP1A
Status: Completed | Type: Observational
Sponsor: Lia Bally (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: DEEP1A
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Bariatric Surgery; Hypoglycemia; Gastric Bypass
Keywords: Insulin turnover; Insulin secretion; Deuterated Water; De-novo insulin synthesis
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHH patients: Patients following Roux-en-Y gastric bypass surgery (≥1 year ago) with confirmed post-prandial hyperinsulinemic hypoglycemia
  Interventions: Other: Heavy water experiment
- Healthy controls: Non-PHH, non-surgical healthy individuals
  Interventions: Other: Heavy water experiment

INTERVENTIONS:
Other: Heavy water experiment — 3 times daily heavy water (deuterated-water) and mixed meal administration for one week

SUMMARY:
The primary objective of this study is to observe the kinetics of pre-stored and de-novo synthesized insulin that is secreted into the circulation using an in-vivo heavy water (D2O) labelling experiment in patients with postprandial hyperinsulinaemic hypoglycaemia (PHH) and non-surgical non-PHH controls.

DETAILED DESCRIPTION:
Despite an increased prevalence, the underlying pathophysiology of PHH remains incompletely understood. It is generally assumed that PHH is caused by excess insulin secretion, either due to an intrinsic beta-cell abnormality (histology showing increased beta-cell mass or signs of hyperfunction) and/or increased postprandial insulinotropic signals (also known as the incretin-effect) as a consequence of the re-arranged gastrointestinal tract and accelerated nutrient transit and absorption. Either of the two explanations would imply an altered insulin turnover in these patients with higher amounts of pre-stored insulin and/or accelerated de-novo insulin synthesis in response to stimulus-depletion of the available insulin pool. A non-invasive in vivo technique to study insulin turnover has not been established yet and data related to PHH are consequently lacking.

The primary objective of this study is to observe the kinetics of pre-stored and de-novo synthesized insulin that is secreted into the circulation using an in-vivo heavy water (D2O) labelling experiment in patients with postprandial hyperinsulinaemic hypoglycaemia (PHH) and non-surgical non-PHH controls. The investigators hypothesize that the suggested methodological approach is feasible to assess insulin turnover and provides the foundation for further studies in different target groups.

ELIGIBILITY:
Inclusion criteria for PHH patients:

* Aged ≥18 years
* Roux-en-Y gastric bypass ≥1 year ago
* PHH defined as postprandial plasma or sensor glucose<3.0mmol/l according to the International Hypoglycaemia Study Group and exclusion of other causes of hypoglycaemia

Inclusion criteria for non-PHH non-surgical controls:

* Aged ≥18 years
* Absence of any condition or previous surgery known to affect gastro-intestinal integrity and food absorption

Exclusion Criteria:

* Clinically relevant weight changes (≥5%) within the past 3 months
* Incapacity to give informant consent
* Historical or current diabetes based on HbA1c ≥6.5% without glucose-lowering treatment
* Haemoglobin level below 13.5 g/l
* Ongoing treatment with glucose-lowering drugs, anorectic drugs, steroids or any medications known to affect gastric motility
* Active heart, lung, liver, gastrointestinal, renal or neurological disease
* Inability to follow study procedures
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by referral from our outpatient endocrine clinic and collaborating Centres of Excellence for Metabolic Surgery. Non-surgical controls will be recruited through advertisement according to guidelines from swissethics.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Total amount of pre-stored insulin secreted | During the 7 days of the heavy water administration period
  Measured using deuterium (2H)-labelled insulin in the plasma

SECONDARY OUTCOMES:
Time course of the increase in 2H-labelled insulin in plasma | During the 7 days of the heavy water administration period
Time course of the increase in 2H-labelled insulin in urine | During the 7 days of the heavy water administration period
Time course of the increase in 2H-labelled c-peptide in plasma | During the 7 days of the heavy water administration period
Time course of the increase in 2H-labelled c-peptide in urine | During the 7 days of the heavy water administration period

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — Bern University Hospital, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No